CLINICAL TRIAL: NCT01675479
Title: A Prospective Study to Evaluate the Safety and Effectiveness of Wavefront-Guided Lasik Correction of Hyperopic Refractive Errors With the iDesign Advanced Wavescan Studio™ System and Star S4 IR™ Excimer Laser System
Brief Title: Safety and Effectiveness of Wavefront-Guided LASIK Correction of Hyperopic Refractive Errors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR-111-IDHP
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Results first posted 2018-04-25 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Hyperopia
Keywords: refractive; errors
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- wavefront-guided LASIK (Experimental)
  Interventions: Device: LASIK correction of hyperopic refractive errors

INTERVENTIONS:
Device: LASIK correction of hyperopic refractive errors — Surgeons will perform wavefront-guided LASIK based upon measurement obtained with the iDesign System

SUMMARY:
Demonstrate that wavefront-guided LASIK using measurements from the iDesign System is safe and effective for the treatment of Hyperopia.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of pre-operative exam
* Best Spectacle Corrected Visual Acuity (BSCVA) of 20/20 or better
* Demonstration of refractive stability
* Anticipated post-operative stromal bed thickness of at least 250 microns
* Willing and capable of returning for follow-up examinations for the duration of the study

Exclusion Criteria:

* Women who are pregnant, breast-feeding, or intend to become pregnant over the course of the study
* Concurrent use of topical or systemic medications that may impair healing
* History of any medical conditions that could affect wound healing
* History of prior intraocular or corneal surgery, active ophthalmic disease, or other ocular abnormality
* Evidence of keratoconus, corneal irregularity, or abnormal topography in the operative eye(s)
* Known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2012-12-31 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (9):
- United States (9):
  - Maloney Vision Institute, Los Angeles, California
  - University of Miami Bascom Palmer Eye Institute, Miami, Florida
  - Kraff Eye Institute, Chicago, Illinois
  - Pepose Vision Institute, Chesterfield, Missouri
  - Durrie Vision, Kansas City, Missouri
  - Coleman Vision, Albuquerque, New Mexico
  - Lehmann Eye Center, Nacogdoches, Texas
  - The Eye Center, Fairfax, Virginia
  - King LASIK, Renton, Washington

IPD SHARING:
Plan to Share IPD: No
No Plan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 167 subjects were consented in the study, of which 69 subjects had one or both eyes treated for a total of 135 treated eyes.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Wavefront-Guided LASIK
Started | 69; 135 eyes
Completed | 58; 112 eyes
Not Completed | 11; 23 eyes
Not completed — Lost to Follow-up | 11

BASELINE CHARACTERISTICS:
Groups:
- Wavefront-Guided LASIK: LASIK : Surgeons will perform wavefront-guided LASIK based upon measurement obtained with the iDesign System for correction of hyperopic refractive errors
Arm/Group | Wavefront-Guided LASIK
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 58
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes With a Loss of >2 Lines for Best Spectacle Corrected Visual Acuity (BSCVA)
Description: Hypothesis: <5% of eyes will have a loss of > 2 lines of BSCVA at any postoperative visit, as measured using ETDRS logMAR visual acuity charts at 4 meters
Time Frame: 12 Months
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Groups:
- Wavefront-Guided LASIK: LASIK : Surgeons performed wavefront-guided LASIK based upon measurement obtained with the iDesign System for correction of hyperopic refractive errors
Arm/Group | Wavefront-Guided LASIK
Number analyzed (Participants) | 67
Number analyzed (eyes) | 131
eyes | 2

2. Secondary Outcome: Number of Eyes With Uncorrected Visual Acuity (VA) of 20/40 or Better
Description: Hypothesis: 85% of eyes will have uncorrected visual acuity of 20/40 or better, as measured using ETDRS logMAR charts at 4 meters
Time Frame: 12 Months
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Wavefront-Guided LASIK
Number analyzed (Participants) | 67
Number analyzed (eyes) | 131
eyes | 123

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Wavefront-Guided LASIK
All-Cause Mortality (participants affected / at risk) | 0/69
Serious Adverse Events (participants affected / at risk) | 3/69
Other Adverse Events (participants affected / at risk) | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Wavefront-Guided LASIK (N=69)
Epithelial ingrowth requiring non refractive intervention (Eye disorders) | 1
Decrease in BSCVA (Eye disorders) | 1
Cataract (Eye disorders) | 1
Severe glare (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communications prior to public release and can embargo communications regarding trial results at any time.